CLINICAL TRIAL: NCT02610790
Title: Evaluation of Pre- and Post-operative Physical Activity on Postoperative Rehabilitation After Colorectal Surgery With a Connected Device
Brief Title: BRacelet And Physical actiVity Evaluation (BRAVE)
Acronym: BRAVE
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Nicolas DEMARTINES, Chief Department, University of Lausanne Hospitals
Other Study IDs: 383/15
Record Dates: First submitted 2015-11-08; First posted 2015-11-20 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity
Keywords: connected bracelets, footsteps
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Connected bracelet: Patients with a colorectal surgery planned will be included. Fifteen days before surgery, patients will have a connected bracelet permitting to quantify the number of steps and distance achieved each day before surgery.

SUMMARY:
The aim of this study is to quantify pre- and postoperative physical activity of patients operated on colorectal surgery. Daily physical activity (No. of footsteps) is going to be recorded from 15 days before surgery to the end of hospitalization after surgery in a prospective cohort of consecutive colorectal patients by use of an attached strap. Then, the investigators will propose physical activity thresholds (adapted to the age, gender and patient comorbidities) to optimize the ERAS protocol (Enhanced Rehabilitation After Surgery). Thus, this analysis will allow the investigators to provide patients with physical rehabilitation programs "a la carte" during a hospitalization for colorectal surgery. Connected bracelets will directly involve patients in their care and rehabilitation.

DETAILED DESCRIPTION:
Connected bracelet will be given to 50 consecutive patients undergone colorectal surgery 15 days before surgery. The investigators will measure pre- and postoperative physical activity. It is an observational activity of patient's physical activity during the perioperative period with no intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a colorectal surgery

Exclusion Criteria:

1. Limitation of linguistic or cognitive abilities, interfering with the understanding of the study protocol
2. Lack of consent of the study form
3. Emergency Surgery
4. stoma closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Pre- and postoperative physical activity | 30 days
  Number of footsteps

SECONDARY OUTCOMES:
Quality of life | 30 days
  score (number between 0 to 10)
Quality of sleep | 30 days
  Score (number between 0 to 10)
Pain | 30 days
  Score (number between 0 to 10)
Fatigue | 30 days
  Score (number between 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DEMARTINES, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Department of Visceral Surgery, University Hospital Center, Lausanne, Switzerland